CLINICAL TRIAL: NCT00675701
Title: A Double Blind, Randomized, Repeat-Dose, Parallel Group Study to Define the ECG Effects of Lixivaptan Using a Clinical and a Supratherapeutic Dose, Compared to Placebo and Moxifloxacin (a Positive Control), in Healthy Adult Men and Women: A Thorough ECG Study
Brief Title: A Study to Define the ECG Effects of Lixivaptan Compared to Placebo and Moxifloxacin in Healthy Adult Men and Women: A Thorough ECG Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CardioKine Inc. (Industry)
Collaborators: Cardiokine Biopharma, LLC (Industry); Biogen (Industry)
Responsible Party: Cardiokine, Ink, Cardiokine Biopharma, LLC
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CK-LX1403
Record Dates: First submitted 2008-05-08; First posted 2008-05-12 (Estimated); Last update posted 2011-06-21 (Estimated); Status verified 2008-11

CONDITIONS: Healthy
Keywords: To determine whether lixivaptan administration at supratherapeutic or therapeutic doses results in the prolongation of the QTc interval.
MeSH Terms: interventions — lixivaptan; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Placebo Comparator): Placebo by mouth
  Interventions: Drug: placebo
- B (Experimental): lixivaptan
  Interventions: Drug: lixivaptan
- C (Active Comparator): moxifloxacin
  Interventions: Drug: moxifloxacin

INTERVENTIONS:
Drug: placebo — capsules
  Arms: A
Drug: lixivaptan — capsules
  Arms: B
Drug: moxifloxacin — tablets
  Arms: C

SUMMARY:
This is a Phase 1, double-blind, randomized, repeat-dose, single -dite, 4-arm parallel group study to define the ECG effect of lixivaptan using a therapeutic and supratherapeutic dose compared to placebo and moxifloxacin (a positive control in healthy adult men and women.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or females, between 18 and 45 years of age, inclusive
2. Body mass index (BMI; see 279HAPPENDIX B) within 18 to 32 kg/m2, inclusive
3. Absence of significant disease as determined by medical history, physical examination, laboratory evaluations, 12-lead ECG, and vital signs (conducted at Screening or on admission to the clinic)
4. Normal 12-lead ECG with no clinically significant abnormalities of rate, rhythm, or conduction (i.e., normal PR interval of 0.12-0.2 sec, normal QRS duration of 0.06-0.1 sec, and a QTc Bazett <440 ms for males or <470 ms for females)
5. Clinical laboratory evaluations (including a serum chemistry panel [fasted at least 8 hours], CBC, and UA) within the reference range for the test laboratory. Laboratory findings outside the normal reference range may be repeated once; The subject may be enrolled if laboratory findings outside the normal reference range are deemed not clinically significant by the investigator
6. Negative test for selected drugs of abuse (280HAPPENDIX A) at Screening and at Check-in
7. Women must be postmenopausal (more than 12 months since last period, verified by FSH and estradiol measurements); surgically sterile (hysterectomy or tubal ligation at least 6 months prior to enrollment); or be using an intrauterine device (including hormone-impregnated devices), or double barrier (i.e. diaphragm plus spermicide) non-hormonal contraceptive therapy for the duration of the study; and must have a negative serum pregnancy test at Screening and Check-in
8. Able to communicate effectively with study personnel
9. Be adequately informed of the nature and risks of the study and able to comprehend and sign an Informed Consent Form (ICF) prior to any study related procedures.

Exclusion Criteria:

1. Known hypersensitivity or allergy to lixivaptan (VPA-985), other vasopressin antagonists, moxifloxacin, or any other fluoroquinolones;
2. Women who are pregnant or breast feeding
3. A first degree relative with Long QT Syndrome or a family history of unexplained sudden death
4. Any history, disease or condition (medical or surgical) which, in the opinion of the investigator, might compromise the hematologic, cardiovascular, pulmonary, renal, gastrointestinal, hepatic, urological, neurological, psychiatric, or central nervous system; or other conditions that might interfere with the absorption, distribution, metabolism, or excretion of study drug, or would place the subject at increased risk
5. History of unexplained syncope
6. History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (appendectomy, hernia repair, and/or cholecystectomy will be allowed)
7. History or presence of an abnormal ECG that, in the Investigator's opinion, is clinically significant
8. Screening systolic blood pressure <90 mmHg or >140 mmHg, and/or diastolic blood pressure >90 mmHg
9. Screening heart rate >90 beats per minute
10. Positive screen for hepatitis B (HBsAg), hepatitis C (anti-HCV), or HIV (anti-HIV)
11. Participation in any other investigational study within 30 days prior to Check-in
12. Any history of alcohol abuse, illicit drug use, significant mental illness, physical dependence to any opioid, or any history of drug abuse or addiction within 6 months prior to Check-in
13. A history of difficulty with donating blood
14. Donation of ≥ 500 mL blood or blood products within 45 days prior to enrollment
15. Receipt of blood products within 2 months prior to Check-in
16. Use of any of the medications in 281HTable 3 within the given timeframe prior to Check-in:

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 298 (Actual)
Dates: Start 2008-05; Primary Completion 2008-09 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Timed-matched, placebo-corrected, changed from Baseline in QTc | 7days

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site 1, Austin, Texas, United States